CLINICAL TRIAL: NCT03795324
Title: Red-fleshed Apple as a Novel Anthocyanin-biofortified Food to Improve Cardiometabolic Risk Factors: Innovation in Crop and Application to Health.
Brief Title: Red-fleshed Apple as a Novel Anthocyanin-biofortified Food to Improve Cardiometabolic Risk Factors.
Acronym: AppleCor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Rovira i Virgili (Other)
Collaborators: Universitat de Lleida (Other); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Rosa Sola, MD, PhD, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AppleCor
Record Dates: First submitted 2018-12-21; First posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: High LDL-cholesterol Levels
Keywords: Anthocyanins; apple; biofortification; cardiometabolic; LDL cholesterol; polyphenols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Redlove Apple (Experimental): Redlove Apple intervention
  This product is a biofortified cultivar apple with anthocyanins.
  Interventions: Other: Redlove Apple intervention
- Green Apple (Experimental): Green Apple intervention
  This product is a common cultivar apple without anthocyanins.
  Interventions: Other: Green Apple intervention
- Aronia Drink (Experimental): Aronia drink intervention
  This product is an infusion of aronia fruit extract rich in anthocyanin.
  Interventions: Other: Aronia drink intervention

INTERVENTIONS:
Other: Redlove Apple intervention — The bioactive compounds present in this product are anthocyanins (50mg per 80g of product).It was a 6 weeks nutritional intervention. Volunteers will eat 80g per day of lyophilized redlove apple.
  Arms: Redlove Apple
Other: Green Apple intervention — It was a 6 weeks nutritional intervention. Volunteers will eat 80g per day of lyophilized green apple.
  Arms: Green Apple
Other: Aronia drink intervention — The bioactive compounds present in this extract are anthocyanins (50mg per 1L of water).It was a 6 weeks nutritional intervention. Volunteers will drink 1L per day of an aronia drink
  Arms: Aronia Drink

SUMMARY:
The primary aim is to evaluate the added health value of the presence of anthocyanins in the redlove apple, versus a green apple with a similar matrix, on cardiometabolic risk, and compare the matrix effect on the bioavailability of anthocyanins, and its effect on cardiometabolic risk factors, in two different products with a similar phenolic and anthocyanin content: the redlove apple and an aronia drink.

DETAILED DESCRIPTION:
The worldwide high prevalence of cardiovascular disease (CVD) requires lifestyle changes and new dietary prevention strategies based on the increased intake of foods rich in bioactive compounds, as they are considered as key mediators in the improvement of CVD risk factors.

Regarding the health impact on anthocyanins in cardiometalic risk factors and CVD, it has been reported that the dietary intake of anthocyanidins, among other classes of flavonoids, is inversely associated with the risk of CVD in both European and US population. A recent systematic review of human randomized controlled trials assessing the impact of anthocyanins on CVD markers concluded that one of the main modulated outcomes is the decrease of serum LDLc. However, diet does not appear to be sufficient to guarantee the necessary intake to obtain the health benefits specified. Due to previous positive results, a new dietetic strategy based on biofortification to enhance the levels of phenolic compounds is proposed in the present project.

The primary aim is to evaluate the added health value of the presence of anthocyanins in the redlove apple, versus a green apple with a similar matrix, on cardiometabolic risk, and compare the matrix effect on the bioavailability of anthocyanins and its effect on cardiometabolic risk factors, in two different products with a similar phenolic and anthocyanin content: the redlove apple and an aronia drink.

Participants will be 120 free-living volunteers (men and women) with high LDL-cholesterol levels (LDL-cholesterol levels ≥115 mg/dl and ≥190 mg/dl) who will be assigned to one of the three arms for 6-week period of dietary treatment. The design of the intervention study is controlled, parallel and randomized. The intervention will combine acute (post-prandial) and chronic effects.

The sample size was computed to be sufficient to detect differences between treatment groups regarding the evolution in time of LDL-cholesterol levels. Justification of chosen sample size is based on assuming a 0.50mmol/l (approximately 15%) post-intervention difference of LDL-cholesterol and a 0.72mmol/l Standard deviation (SD), with α=0.05 and 1-β=0.08 a minimum of 22 participants were required. However the sample size will be 40 participants for arm, in total 120 subjects.

For the acute study, the investigators have chosen n=10 subjects per arm according to the most studies that have addressed the metabolic effects of a postprandial intervention have been performed using a very similar number of subjects with statistically good quality results.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* LDL-cholesterol levels ≥115 mg/dl and ≥190 mg/dl.
* Sign the informed consent provided before the initial screening visit.

Exclusion Criteria:

* LDL-cholesterol levels ≤115 mg/dl and <190 mg/dl.
* Use of hypolipemiant treatment (drugs and functional foods), or hypoglucaemiant treatment.
* Having diabetes mellitus type 1 or type 2.
* BMI values ≥35kg/m2.
* Present triglycerides levels ≥350mg/dl.
* Presenting anemia (hemoglobin ≤13g/dl in men and ≤12g/dl in women).
* Subjects diagnosed of intestinal disorders such as Chron disease, colitis ulcerous, celiac disease and irritable bowel syndrome.
* Present fructose and/or sorbitol and/or gluten intolerance.
* Present clinical active chronic disease
* Use of antioxidants supplements.
* Being pregnant or intending to become pregnant.
* Be in breastfeeding period.
* Present chronic alcoholism.
* Tobacco use.
* Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
* Being unable to follow the study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Changes in serum LDL-cholesterol (measured in mg/dL) | 6 weeks, week 1 and week 6
  Serum lipids will be measured by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland). Then, LDL-cholesterol will be alculated by the Friedewald formula.

SECONDARY OUTCOMES:
Changes in parameters of body composition (weight measured in kg) | 6 weeks, week 1, week 2, week 4 and week 6
  Trained dieticians measure weight using a body composition analyzer (Tanita SC 330-S; Tanita Corp., Barcelona, Sapin)
Parameters of body composition (height measured in meters) | 6 weeks, week 1
  Trained dieticians measure height using a well mounted stadiometer (Tanita Leicester Portable; Tanita Corp., Barcelona, Spain).
Changes in parameters of body composition (BMI measured in kg/m2) | 6 weeks, week 1, week 2, week 4 and week 6
  Body mass index (BMI) is calculated as the ratio between measured weight (kg)/and the square of height (m).
Changes in parameters of body composition (waist circumference measured in cm) | 6 weeks, week 1, week 2, week 4 and week 6
  Waist circumference (WC) is measured at the umbilicus using a 150 cm anthropometric steel measuring tape.
Changes in blood pressure (systolic blood pressure and diastolic blood pressure measured in mmHg) | 6 weeks, week 1, week 2, week 4 and week 6
  Systolic and diastolic blood pressure (SBP and DBP) are measured twice after 2-5 minutes of patient seated, with one-minute interval in between, using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Changes in ischemic reactive hyperemia (IRH measured in perfusion units) | 6 weeks, week 1 and week 6
  The endothelial-dependent vasomotor functions will be measured as IRH by a Laser-Doppler linear Periflux 5000 flowmeter (Perimed AB, Järfälla, Stockholm, Sweden)
Changes in lipid plasmatic markers (total cholesterol, HDL cholesterol, triglycerides, non-esterified fatty acids, Apo B100 and Apo A. All these lipid plasmatic markers will be measured in mg/dL) | 6 weeks, week 1 and week 6
  Total cholesterol, HDL cholesterol, triglycerides, non-esterified fatty acids, Apo B100 and Apo A will be measured by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland).
Changes in glucose markers (glucose and insulin measured in mg/dL) | 6 weeks, week 1 and week 6
  measured by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland).
Changes in oxidative markers (LDLox and Endogenous fat soluble antioxidants measured in mg/dL) | 6 weeks, week 1 and week 6
  Plasma oxidized LDL measured by ELISA kit (Mercodia AB, Uppsala, Sweden). The analysis of fat-soluble vitamins (vitamin D, alpha-tocopherol, and carotenoids) will be carried out in whole blood with DBS cards. The determinations will be performed by ultra-performance liquid chromatography (UPLC) coupled to photodiode array (PDA) and tandem mass spectrometry (MS/MS) detectors.
Changes in inflammation markers (c-reactive protein and serum endothelin-1 measured in mg/dL) | 6 weeks, week 1 and week 6
  Serum high sensitive C reactive measured by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Serum endothelin type 1 measured by ELISA kits (R&D Systems, Minneapolis, USA).
Changes in dietary compliance markers (Phenolic compounds and metabolites measured in mg/L in 24h urine samples) | 6 weeks, week 1 and week 6
  will be analysed by UPLC-MS/MS as previously described.
Changes in faeces metabolites (Short Chain Fatty Acids, bile acids and sterols measured in mg/L in faeces samples) | 6 weeks, week 1 and week 6
  will be performed by gas chromatography (GC).
Changes in fecal microbiota composition (relative abundance of the identified operational taxonomic units (OTUs) measured as % change from baseline) | 6 weeks, week 1 and week 6
  will be studied by sequencing its whole genomic content. Illumina platform will be used to obtain the metagenomics and metatranscriptomics of each sample following previous protocols developed.
Changes in lipoprotein profile (number of LDL and HDL particles measured as % change from baseline) | 6 weeks, week 1 and week 6
  Number of particles and size LDL and HDL measured by NMR technology, in a Vantera Clinical Analyzer (LipoScience Inc., Raleigh, NC, USA).
Changes in cholesterol efflux (measured as % change from baseline) | 6 weeks, week 1 and week 6
  Cholesterol efflux measured by in vitro assays in Murine J-774A.1 macrophages labeled with TopFluor-Cholesterol, a fluorescent cholesterol probe in which the cholesterol molecule is linked to boron dipyrromethene difluoride (BODIPY) moiety (Avanti Polar Lipids, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Sola, MD, PhD, Principal Investigator — University Rovira i Virgili
Locations (1):
- University Rovira i Virgili, Reus, Tarragona, Spain

REFERENCES:
- [Derived] Macia A, Romero MP, Pedret A, Sola R, Clifford MN, Rubio-Pique L. Assessment of human inter-individual variability of phloretin metabolites in urine after apple consumption. AppleCOR study. Food Funct. 2023 Nov 27;14(23):10387-10400. doi: 10.1039/d3fo02985a. PMID 37933196